CLINICAL TRIAL: NCT06083532
Title: The Effect of Post-activation Potentiation on Lower Limb Explosive Force in Collegiate Male Basketball Players in China
Brief Title: Effect of PAP on Lower Limb Explosive Force in Basketball Players in CHINA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Jiazhe Li, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Li Jiazhe
Record Dates: First submitted 2023-10-02; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Physical Fitness
Keywords: post-activation potentiation; lower limbs explosive force; complex training; male basketball players; dynamic warm-up

STUDY DESIGN:
Intervention Model Description: In this experiment, the experimental group conducted the post-activation potentiation combined with complex training content intervention designed in this study. In contrast, the control group will perform a training program that combines warm-up routine methods with complex training.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PAP induced at an intensity of 70% 1RM（One-Repetition Maximum）combined with complex training (Experimental): PAP induced at an intensity of 70% 1RM combined with complex training was shown over the 12 weeks.
  Interventions: Behavioral: PAP induced at an intensity of 70% 1RM combined with complex training
- PAP induced at an intensity of 80% 1RM combined with complex training (Experimental): PAP induced at an intensity of 80% 1RM combined with complex training was shown over the 12 weeks.
  Interventions: Behavioral: PAP induced at an intensity of 80% 1RM combined with complex training
- PAP induced at an intensity of 90% 1RM combined with complex training (Experimental): PAP induced at an intensity of 90% 1RM combined with complex training was shown over the 12 weeks.
  Interventions: Behavioral: PAP induced at an intensity of 90% 1RM combined with complex training
- Routine warm-up combined with complex training (Active Comparator): Routine warm-up combined with complex training was shown over the 12 weeks.
  Interventions: Behavioral: Routine warm-up combined with complex training

INTERVENTIONS:
Behavioral: PAP induced at an intensity of 70% 1RM combined with complex training — This group of subjects first performed 3 sets of 70% 1RM squats after a routine warm-up, 3 times per set, with an interval of 2 minutes between sets. The entire process was maintained for 30 minutes, and then after a 6-minute rest, they performed complex training consists of maximum strength training (back squats) and plyometric training (drop Jump). The Intensity & Repetition of back squats is 80% 1RM × 4, 4 sets, interval time is 2min; rest for 3 minutes. , perform drop jump, intensity & repetition is 50cm (height) × 10, 4 sets, and the rest time is 2 minutes. Intervention training was conducted twice weekly for 12 weeks,and the intensity is gradually increasing over the 12 weeks.
  Arms: PAP induced at an intensity of 70% 1RM（One-Repetition Maximum）combined with complex training
Behavioral: PAP induced at an intensity of 80% 1RM combined with complex training — This group of subjects first performed 3 sets of 80% 1RM squats after a routine warm-up, 2 times per set, with an interval of 2 minutes between sets. The entire process was maintained for 30 minutes, and then after a 6-minute rest, they performed complex training consists of maximum strength training (back squats) and plyometric training (drop Jump). The Intensity & Repetition of back squats is 80% 1RM × 4, 4 sets, interval time is 2min; rest for 3 minutes. , perform drop jump, intensity & repetition is 50cm (height) × 10, 4 sets, and the rest time is 2 minutes. Intervention training was conducted twice weekly for 12 weeks,and the intensity is gradually increasing over the 12 weeks.
  Arms: PAP induced at an intensity of 80% 1RM combined with complex training
Behavioral: PAP induced at an intensity of 90% 1RM combined with complex training — This group of subjects first performed 3 sets of 90% 1RM squats after a routine warm-up, 1 times per set, with an interval of 2 minutes between sets. The entire process was maintained for 30 minutes, and then after a 6-minute rest, they performed complex training consists of maximum strength training (back squats) and plyometric training (drop Jump). The Intensity & Repetition of back squats is 80% 1RM × 4, 4 sets, interval time is 2min; rest for 3 minutes. , perform drop jump, intensity & repetition is 50cm (height) × 10, 4 sets, and the rest time is 2 minutes. Intervention training was conducted twice weekly for 12 weeks,and the intensity is gradually increasing over the 12 weeks.
  Arms: PAP induced at an intensity of 90% 1RM combined with complex training
Behavioral: Routine warm-up combined with complex training — This group of subjects first completed a 30-minute routine warm-up, then rested for 6 minutes, and then performed complex training consisted of maximum strength training (back squats) and plyometric training (drop jump). Back squat intensity & repetition is 80% 1RM × 4, 4 sets, with an interval of 2 minutes; after resting for 3 minutes, perform a drop jump, Intensity & Repetition is 50cm (height) × 10, 4 sets, with an interval of 2 minutes. Intervention training was conducted twice weekly for 12 weeks, and the intensity was gradually increasing over the 12 weeks.
  Arms: Routine warm-up combined with complex training

SUMMARY:
The phenomenon that high-intensity warm-up activities help improve muscle strength and explosive performance is called post-activation potentiation (PAP), which is a warm-up method that uses high-intensity stimulation to induce the activation of more type II muscle fibers. However, the results of studies exploring the enhancing effect of PAP on lower limb explosive strength are still controversial. In studies with no significant difference, it is believed that there are many factors that affect PAP, such as activation method, activation intensity, recovery time and individual factors, etc., and it is difficult to control during implementation. In addition, traditional warm-up methods such as jogging and stretching have been shown to have limited effectiveness in improving athletes' performance. In the past, there have been many studies on the combination of PAP and lower limb explosive strength, but there are almost no studies on the long-term effects of PAP on the lower limb explosive strength of basketball players. Therefore, this study studies the characteristics of PAP in order to find the best activation scheme for PAP, and then combines the enhancement effect of PAP with the explosive power of the lower limbs to improve the explosive power of the lower limbs of basketball players, and verifies the long-term effect of combining PAP with explosive power training. In order to provide new changes and breakthroughs in the design of physical training for basketball players and improve the sports performance of college male basketball players.

DETAILED DESCRIPTION:
The study was a four-groups randomized controlled trial. In the study, the experimental group conducted a 12-week post-activation potentiation combined with lower limb explosive training intervention designed in this study. In contrast, the control group also underwent a 12-week lower limb explosive training intervention, but the warm-up method was conventional warm-up activities. Subjects participated in training intervention programs twice weekly. After the 12-week training program, data collection was completed.

1. Warm-up content： The experimental group used PAP as a warm-up method and performed pre-stimulation to induce post-activation potentiation. The pre-activation method is back squats. The pre-activation intensity and frequency are 70% 1RM （One-Repetition Maximum） × 3, 80% 1RM × 2, 90% 1RM × 1 respectively, and the interval time is 2 minutes. The control group performed routine warm-up activities.
2. Explosive strength training content for lower limbs： After completing the warm-up activities, there was a six-minute interval, and then the experimental group and the control group began the same explosive training content of the lower limbs.

ELIGIBILITY:
Inclusion Criteria:

* The population must be collegiate male basketball players and between the ages of 18 and 22；
* Contestants must be in good health, and must have a physical training background；
* Only students who can complete these training requirements can be included in the research data.

Exclusion Criteria:

* Collegiate female basketball players should be excluded from this study;
* Players with less than one year of physical training experience;
* Participants were not healthy collegiate male basketball players such as injured players, mental patient or special students who were seriously depressed, sub-health;
* Students who are consistently late or absent from training sessions will eventually be excluded.

Ages: 18 Years to 22 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-01-20 (Estimated); Study Completion 2024-02-15 (Estimated)

PRIMARY OUTCOMES:
Counter Movement Jump performance of subjects （height） | Pre-test: Before experiment; Post-test: 12 weeks end.
  This indicator is used to test the explosive force of the lower body. And by measuring it, we can get its jump height, Rate of Force Development, the Peak Rate Force Development, Peak Power, the Peak Ground Vertical Reaction Force, which are used to analyze the changes in the explosive force of the lower limbs in detail.
Drop Jump performance of subjects （height） | Pretest: Before experiment; Post-test: 12 weeks end.
  This indicator is used to test the explosive force of the lower body. And by measuring it, we can get its jump height, Rate of Force Development, the Peak Rate Force Development, Peak Power, the Peak Ground Vertical Reaction Force, which are used to analyze the changes in the explosive force of the lower limbs in detail.
Squat Jump performance of subjects （height） | Pre-test: Before experiment; Post-test: 12 weeks end.
  This indicator is used to test the explosive force of the lower body. And by measuring it, we can get its jump height, Rate of Force Development, the Peak Rate Force Development, Peak Power, the Peak Ground Vertical Reaction Force, which are used to analyze the changes in the explosive force of the lower limbs in detail.
Run-up right-foot take-off, Run-up left-foot take-off performance of subjects（height） | Pre-test: Before experiment; Post-test: 12 weeks end.
  This indicator is used to test the explosive force of the lower body. And by measuring it, we can get its jump height, Rate of Force Development, the Peak Rate Force Development, Peak Power, the Peak Ground Vertical Reaction Force, which are used to analyze the changes in the explosive force of the lower limbs in detail.
30-meter sprint performance of subjects（time） | Pre-test: Before experiment; Post-test: 12 weeks end.
  By testing the subject's 30-meter sprint time, changes in the explosive power of the lower limbs can be observed.

CONTACTS AND LOCATIONS:
Overall Officials: Jiazhe Li, PhD, Principal Investigator — Universiti Putra Malaysia
Locations (1):
- Wuhan Sports University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
Since this is my doctoral thesis experiment, I won't share it until I graduate.

REFERENCES:
- [Result] Golas A, Maszczyk A, Zajac A, Mikolajec K, Stastny P. Optimizing post activation potentiation for explosive activities in competitive sports. J Hum Kinet. 2016 Sep 10;52:95-106. doi: 10.1515/hukin-2015-0197. eCollection 2016 Sep 1. PMID 28149397
- [Result] Kobal R, Pereira LA, Kitamura K, Paulo AC, Ramos HA, Carmo EC, Roschel H, Tricoli V, Bishop C, Loturco I. Post-Activation Potentiation: Is there an Optimal Training Volume and Intensity to Induce Improvements in Vertical Jump Ability in Highly-Trained Subjects? J Hum Kinet. 2019 Oct 18;69:239-247. doi: 10.2478/hukin-2019-0016. eCollection 2019 Oct. PMID 31666906
- [Result] Kilduff LP, Owen N, Bevan H, Bennett M, Kingsley MI, Cunningham D. Influence of recovery time on post-activation potentiation in professional rugby players. J Sports Sci. 2008 Jun;26(8):795-802. doi: 10.1080/02640410701784517. PMID 18569545
- See also: This article is from National Library of Medicine — http://pubmed.ncbi.nlm.nih.gov/28149397/
- See also: This article is from National Library of Medicine — http://pubmed.ncbi.nlm.nih.gov/31666906/
- See also: This article is from National Library of Medicine — http://pubmed.ncbi.nlm.nih.gov/18569545/